CLINICAL TRIAL: NCT06120842
Title: A Prospective, Multicenter, Randomized, Masked, Controlled Study to Evaluate the Safety, Efficacy, and Dose-response of the Bimatoprost Implant System Used in Combination With the SpyGlass IOL Compared to Timolol Maleate Ophthalmic Solution, USP, 0.5%
Brief Title: Evaluation of the Bimatoprost Implant System Used in Combination With the SpyGlass Intraocular Lens Compared to Timolol Ophthalmic Solution
Acronym: Tigris
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SpyGlass Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGP-003
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cataract; Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Cataract; Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Bimatoprost Implant System (High Dose) / IOL Combination (Experimental)
  Interventions: Drug: Bimatoprost Implant System (High Dose); Device: SpyGlass IOL
- Bimatoprost Implant System (Low Dose) / IOL Combination (Experimental)
  Interventions: Drug: Bimatoprost Implant System (Low Dose); Device: SpyGlass IOL
- Timolol Maleate Ophthalmic Solution 0.5% (Active Comparator)
  Interventions: Drug: Timolol Maleate Ophthalmic Solution, 0.5%; Device: Commercially Available Aspheric Monofocal Non-Yellow Chromophore IOL

INTERVENTIONS:
Drug: Bimatoprost Implant System (High Dose) — Bimatoprost Implant System (High Dose) used in combination with the SpyGlass IOL
  Arms: Bimatoprost Implant System (High Dose) / IOL Combination
Drug: Bimatoprost Implant System (Low Dose) — Bimatoprost Implant System (Low Dose) used in combination with the SpyGlass IOL
  Arms: Bimatoprost Implant System (Low Dose) / IOL Combination
Drug: Timolol Maleate Ophthalmic Solution, 0.5% — Timolol Maleate Ophthalmic Solution 0.5% BID
  Arms: Timolol Maleate Ophthalmic Solution 0.5%
Device: Commercially Available Aspheric Monofocal Non-Yellow Chromophore IOL — Commercially Available Aspheric Monofocal Non-Yellow Chromophore Intraocular Lens
  Arms: Timolol Maleate Ophthalmic Solution 0.5%
Device: SpyGlass IOL — SpyGlass Intraocular Lens
  Arms: Bimatoprost Implant System (High Dose) / IOL Combination; Bimatoprost Implant System (Low Dose) / IOL Combination

SUMMARY:
This trial is a randomized study to evaluate and compare two doses of the Bimatoprost Implant System used in combination with the SpyGlass IOL to Timolol Ophthalmic Solution in participants with mild to moderate open-angle glaucoma or ocular hypertension undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate open-angle glaucoma or ocular hypertension
* Planned removal of cataract
* Female participants of childbearing potential must have a negative urine pregnancy test at the baseline visit and agree to the use of contraception

Exclusion Criteria:

* Uncontrolled systemic disease
* History of incisional/refractive corneal surgery
* Any glaucoma diagnosis other than OHT, open-angle, pseudoexfoliation, or pigmentary glaucoma
* History of incisional glaucoma surgery or intraocular injections
* Other ocular diseases, pathology, or conditions

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Mean IOP Reduction from Baseline (mmHg) | Weeks 2 and 6, and Month 3
  Time matched mean IOP reduction from Baseline (mmHg) in the study eyes at all the individual IOP timepoints

SECONDARY OUTCOMES:
Mean IOP | Weeks 2 and 6 and Months 3, 6, 12, 18, 24, 27, 30, 33, and 36
  Time matched mean IOP (mmHg) at Weeks 2 and 6 and Months 3, 6, 12, 18, 24, 27, 30, 33, and 36
Mean IOP Change from Baseline | Months 6, 12, 18, 24, 27, 30, 33, and 36
  Time matched mean IOP change from Baseline (mmHg) at Months 6, 12, 18, 24, 27, 30, 33, and 36
Time to postoperative introduction of IOP-lowering medications | Total Study Period of 36 Months
  Time (Days) to postoperative introduction of IOP-lowering medications (IOP-lowering medications other than the study treatments)
Number of IOP-lowering medications introduced postoperatively | Total Study Period of 36 Months
  Number of IOP-lowering medications introduced postoperatively (N) at Weeks 2 and 6, and Months 3, 6, 12, 18, 24, 27, 30, 33, and 36
Proportion of eyes achieving BCDVA 20/40 or better | Months 3, 6, and 12
  Snellen Equivalent
Manifest refraction spherical equivalent | Month 3
  Manifest refraction spherical equivalent (MRSE)

OTHER OUTCOMES:
Number and Rates of Adverse Events | Total Study Period of 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hafner, Study Chair — SpyGlass Pharma, Inc.
Locations (1):
- Arizona Advanced Eye Research Institute, Glendale, Arizona, United States

REFERENCES:
- See also: SpyGlass Pharma Website — https://www.spyglasspharma.com/